CLINICAL TRIAL: NCT02302365
Title: Multicenter, Retrospective Data Collection of Routine Clinical Use With the Spectra Optia® Apheresis System for White Blood Cell Depletion
Brief Title: Data Collection of Routine Clinical Use With the Spectra Optia® Apheresis System for White Blood Cell Depletion
Acronym: WBCD
Status: Completed | Type: Observational
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Other Study IDs: CTS-5043
Record Dates: First submitted 2014-11-18; First posted 2014-11-27 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Leukocytosis
Keywords: white blood cell depletion; apheresis
MeSH Terms: conditions — Leukocytosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spectra Optia® Apheresis System — White Blood Cell Depletion

SUMMARY:
This study is a multicenter, retrospective data collection of routine clinical use with the Spectra Optia® apheresis system for white blood cell depletion.

DETAILED DESCRIPTION:
The goal of this study is to gather a broader knowledge and information from routine clinical use on the performance and safety of white blood cell depletion procedures with the Spectra Optia® apheresis system.

In order to do so, retrospective data on white blood cell depletion procedures with the Spectra Optia® apheresis system done in routine use in 3 different centers will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received a minimum of 1 white blood cell depletion procedure via the Spectra Optia Apheresis System

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone white blood cell depletion via the Spectra Optia Apheresis System which is likely to include patients with severe leukocytosis in acute leukemia (acute myeloid leukemia, acute lymphoblastic leukemia, or in chronic myelogenous leukemia) or to prevent tumor lysis syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isobelle Galeon, MD, MPH, MSCS, Study Director — Medical Monitor, Clinical Safety
Locations (3):
- UZ Gasthuisberg, Leuven, Belgium
- Institute for Transfusion Medicine and Immunohaematology, German Red Cross Blood Donor Service Baden-Württemberg-Hessen gGmbH, Johann-Wolfgang-Goethe-University Hospital, Frankfurt am Main, Germany
- Szent Istvan and Szent Laszlo Hospital of Budapest, Budapest, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Who Received a Minimum of 1 WBCD Procedure: Eligible subjects had received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System
Period: 0-2 Hour Period
Arm/Group | Subjects Who Received a Minimum of 1 WBCD Procedure
Started | 43 (Data were collected from 58 WBCD procedures performed in 43 subjects - Full and Safety Analysis Sets)
Completed | 41 (The Per-protocol Analysis Set comprised 54 procedures performed in 41 subjects)
Not Completed | 2
Period: 0-24 Hour Period
Arm/Group | Subjects Who Received a Minimum of 1 WBCD Procedure
Started | 32 (2 of 3 study sites collected additional safety data; 32 pts. 0-24 hour data, 43 pts. 0-2 hour data)
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible subjects had received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System.
Groups:
- Subjects Who Received At Least 1 WBCD Apheresis Procedure: Eligible subjects who received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System
Arm/Group | Subjects Who Received At Least 1 WBCD Apheresis Procedure
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 9
  Germany | 11
  Hungary | 23
Weight [Mean (Standard Deviation); unit: kg] | 73.2 (16.7)
Height [Mean (Standard Deviation); unit: cm] | 170.9 (10.3)
Total Blood Volume [Mean (Standard Deviation); unit: Liters] | 4.7 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Decrease in White Blood Cell Count in Patient Following Apheresis Procedure
Description: Percent decrease in WBC count calculation: (WBCpre - WBCpost) / WBCpre x 100%
Time Frame: immediately after apheresis procedure: on average this will be within 15 minutes after the end of the procedure
Population: The Full Analysis Set comprised all 43 patients (58 procedures) for whom WBCD data were collected. One patient terminated the first procedure prematurely and therefore did not have post-procedure data, resulting in a total of 57 units analyzed.
Measure: Mean (Standard Deviation); unit: % change in subject's WBC count
Units Other Than Participants: procedures
Groups:
- WBCD Procedures Performed: Eligible subjects received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System; 58 WBCD procedures were performed in 43 patients
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 57
% change in subject's WBC count | 54.5 (21.40)

2. Primary Outcome: Collection Efficiency (CE) for WBC (or Percent of Processed WBCs) Achieved by Spectra Optia.
Description: Collection efficiency for WBC achieved by Spectra Optia System calculation: (WBC/µL depletion product x depletion product volume) / (WBCpre + WBCpost) / 2 x total processed blood volume)
Time Frame: immediately after apheresis procedure: on average this will be within 15 minutes after the end of the procedure
Population: The CE of the WBCD procedures was measured from the waste bag (depletion product) contents from Sites 2 and 3. WBC counts were not available from the waste bags for subjects treated at Site 1.
Measure: Mean (Standard Deviation); unit: percent of processed WBCs
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 34
Number analyzed (procedures) | 43
percent of processed WBCs | 58.7 (16.1)

3. Primary Outcome: Adverse Events
Description: Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medical device, whether or not considered related to the medical device and/or procedure. Therefore, an AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the medical device and/or procedure.
Time Frame: Participants were followed for the duration of the procedure and for up to 24 hours after the procedure.
Population: Full and Safety Analysis Sets. 53.5% of subjects with acute myeloid leukemia (AML), 18.6% of subjects with chronic lymphocytic leukemia, < 10% of subjects with other diagnoses. The WBCD procedure was performed most frequently to treat leukocytosis (44.2%), to prevent tumor lysis syndrome (34.9%), or to treat increased blood viscosity (20.9%).
Measure: Number; unit: Number of subjects with at least 1 TEAE
Groups:
- Safety Data Collection 0-2 Hours Post Apheresis Procedure: 58 WBCD procedures were performed in 43 patients. Safety data was collected for up to 2 hours post apheresis procedure
- Safety Data Collection 0-24 Hours Post Apheresis Procedure: 41 WBCD procedures were performed in 32 patients. Safety data was collected for up to 24 hours post apheresis procedure
Arm/Group | Safety Data Collection 0-2 Hours Post Apheresis Procedure | Safety Data Collection 0-24 Hours Post Apheresis Procedure
Number analyzed (Participants) | 43 | 32
Number of subjects with at least 1 TEAE | 37 | 30

4. Other Pre Specified Outcome: Pre-procedure WBC Count
Description: Pre-procedure WBC count
Time Frame: Prior to Each Spectra Optia Apheresis Procedure
Population: The Full Analysis Set comprised all 43 patients (58 procedures) for whom WBCD data were collected.
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Units Other Than Participants: procedures
Groups:
- WBCD Procedures Performed: 58 WBCD procedures were performed in 43 patients.
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
cells x 10^9/L | 243.5 (175.6)

5. Other Pre Specified Outcome: Post-procedure WBC Count
Description: Post-procedure WBC count
Time Frame: Following apheresis procedure
Population: Data were collected on a total of 58 procedures, however one patient terminated the first procedure prematurely and therefore did not have post-procedure data.
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Units Other Than Participants: procedure
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedure) | 57
cells x 10^9/L | 119.9 (156.05)

6. Other Pre Specified Outcome: Patient's Platelet Count Pre-depletion Procedure
Description: Patient's platelet count pre-depletion procedure
Time Frame: Prior to Each Spectra Optia Apheresis Procedure
Population: Full and Safety Analysis Sets.
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
cells x 10^3/L | 88.1 (75.58)

7. Other Pre Specified Outcome: Patient's Platelet Count Post-depletion Procedure
Description: Patient's platelet count post-depletion procedure
Time Frame: Participants were followed for the duration of the procedure and for up to 2 hours after the procedure, an average of 6 hours.
Population: Full and Safety Analysis Sets. Data were collected on a total of 58 procedures, however one patient terminated her first procedure prematurely and therefore did not have post-procedure data.
Measure: Mean (Standard Deviation); unit: cells x 10^3/L
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 57
cells x 10^3/L | 59.5 (53.50)

8. Other Pre Specified Outcome: Whole Blood Processed (mL)
Description: Volume of patient's blood processed in mL during the apheresis procedure
Time Frame: as for outcome 7
Population: Full and Safety Analysis Sets
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
mL | 11395 (4010)

9. Post Hoc Outcome: Total Blood Volumes (TBV) Processed
Description: Number of times the patient's TBV was processed during the apheresis procedure based on the patient's estimated TBV (Estimated by Nadler's formula for total blood volume of a human being based on gender, height, and weight).
Time Frame: Post each Spectra Optia Apheresis Procedure
Population: Full and Safety Analysis Sets
Measure: Mean (Standard Deviation); unit: TBV
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
TBV | 2.5 (0.9)

10. Other Pre Specified Outcome: Whole Blood Flow mL/Min
Description: Whole Blood Flow in mL/min measured during the white blood cell depletion procedure
Time Frame: as for outcome 7
Population: Full and Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mL/min
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
mL/min | 50.3 (12.8)

11. Other Pre Specified Outcome: Procedure Duration
Description: The duration of the WBCD procedure measured in minutes
Time Frame: as for outcome 7
Population: Full and Safety Analysis Sets
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 58
minutes | 237.3 (97.38)

12. Other Pre Specified Outcome: Platelet Change (% Change)
Description: % change in patient's pre and post-depletion procedure platelet counts
Time Frame: as for outcome 7
Population: Data were collected on a total of 58 procedures, however one patient terminated her first procedure prematurely and therefore did not have post-procedure data.
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 57
percent change | 20.8 (62.15)

13. Other Pre Specified Outcome: Waste Bag Volume
Description: Volume of the depletion product
Time Frame: Post each Spectra Optia Apheresis Procedure
Population: Full and Safety Analysis Sets; One patient terminated the first procedure prematurely, resulting in a total of 57 units analyzed.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: procedures
Arm/Group | WBCD Procedures Performed
Number analyzed (Participants) | 43
Number analyzed (procedures) | 57
mL | 1371.2 (896.20)

ADVERSE EVENTS:
Time Frame: Adverse event data (including serious adverse events [SAEs]) were collected from the time of the start of the WBCD procedure through 2 hours post-procedure for 43 patients and 58 procedures. Adverse event data (including serious adverse events [SAEs]) were collected from the time of the start of the WBCD procedure through 24 hours post-procedure for 32 patients and 41 procedures.
Description: Adverse events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, and coded using the Medical Dictionary for Regulatory Activities (MedDRA®, version 17.0).
Groups:
- 0-2 Hour Safety Data Collection: Eligible subjects had received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System; safety data collected for 2 hours post apheresis procedure
- 0-24 Hour Safety Data Collection: Eligible subjects had received a minimum of 1 WBCD procedure using the Spectra Optia Apheresis System; safety data collected for 24 hours post apheresis procedure
Arm/Group | 0-2 Hour Safety Data Collection | 0-24 Hour Safety Data Collection
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/32
Other Adverse Events (participants affected / at risk) | 37/43 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0-2 Hour Safety Data Collection (N=43) | 0-24 Hour Safety Data Collection (N=32)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0-2 Hour Safety Data Collection (N=43) | 0-24 Hour Safety Data Collection (N=32)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 19
Anaemia (Blood and lymphatic system disorders) | 15 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 14
Platelet count decreased (Investigations) | 12 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 14
Coagulopathy (Blood and lymphatic system disorders) | 2 | 3
Fatigue (General disorders) | 1 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Hypogammaglobulinaemia (Immune system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Site reserves the right to publish the results of its work on the Study. The timing of publication however shall not exceed the 6 months after completion of the Study. Study Site and the PI agree to submit copies of any manuscript/abstract proposed for publication to Sponsor at least 30 days in advance of the presentation. Sponsor may require the delay of publication for no longer than 90 days for the purpose of filing patent applications.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT02302365/SAP_000.pdf
  • Study Protocol (2014-02-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT02302365/Prot_001.pdf